CLINICAL TRIAL: NCT03172910
Title: Phase 2 Placebo-Controlled, Single-Site, Single-Blind Study of Rivaroxaban Reversal by Ciraparantag as Measured by WBCT
Brief Title: Phase 2 Study of Rivaroxaban Reversal by Ciraparantag as Measured by WBCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PER977-02-012
Record Dates: First submitted 2017-05-19; First posted 2017-06-01 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: PER977; Ciraparantag; Whole Blood Clotting Time (WBCT); Rivaroxaban
MeSH Terms: interventions — PER977; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): ciraparantag (60 mg)
  Interventions: Drug: Ciraparantag; Drug: Rivaroxaban
- Cohort 2 (Experimental): ciraparantag (120 mg)
  Interventions: Drug: Ciraparantag; Drug: Rivaroxaban
- Cohort 3 (Experimental): ciraparantag (180 mg)
  Interventions: Drug: Ciraparantag; Drug: Rivaroxaban
- Cohort 4 (Experimental): ciraparantag (30 mg)
  Interventions: Drug: Ciraparantag; Drug: Rivaroxaban
- Placebo (Placebo Comparator): placebo (saline for injection)
  Interventions: Drug: Placebo; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Ciraparantag — Ciraparantag (administered over 10 minutes)
  Other Names: PER977; AMAG 977
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Placebo — Saline for injection
  Other Names: PBO
  Arms: Placebo
Drug: Rivaroxaban — Rivaroxaban 20 mg given once per day (QD) in the morning

SUMMARY:
This study is a randomized, single-blind, placebo-controlled study to assess the efficacy and safety of ciraparantag administered to healthy volunteers anticoagulated with rivaroxaban measuring clotting times using Whole Blood Clotting Time (WBCT).

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled assessment of the efficacy and safety of ciraparantag administered to healthy volunteers measuring clotting times using WBCT as determined by the manual testing method. All subjects will undergo screening up to 36 days prior to enrollment.

All enrolled subjects are to receive a single dose of 20 mg rivaroxaban in the morning on Days 1-3. On Day 3 (3.75 hours post rivaroxaban), subjects who have a minimum increase in clotting time of 25% (as measured by WBCT) are randomized and will receive a single IV dose 4 hours after the rivaroxaban dose, followed by serial testing of manual WBCT.

Subjects are enrolled sequentially in up to 4 ciraparantag dose cohorts. There will be a safety review after completion of treatment in one cohort and prior to initiation of treatment in the subsequent cohort.

ELIGIBILITY:
General Inclusion Criteria:

1. Adults age 50 to 75 years
2. Laboratory tests (chemistry, hematology and coagulation assessments) and urinalysis performed during screening up to 36 days prior to administration of study treatment deemed not clinically significant by the principal investigator.
3. No clinically significant findings on 12-lead electrocardiogram (ECG) performed during screening
4. Body mass index (BMI) 18 to ≤ 32 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception in addition to their partner using an acceptable form of contraception, when engaging in sexual activity during the course of the study. Moreover, male subjects should not donate sperm or attempt to impregnate a partner during the course of the study and for a period of 12 weeks following discharge from the study.
6. Female subjects must have a negative urine pregnancy test at screening AND: be surgically sterile OR postmenopausal for the last three months, OR in a monogamous relation with a male partner who has undergone a documented vasectomy a minimum of 6 months prior to study commencement. All females must agree to continue to use their method of birth control for the duration of the study and for a minimum of one complete menstrual cycle or 28 days following discharge from the study
7. Subjects who have participated in a prior study of ciraparantag must have been discharged from the study a minimum of 1 month prior to the planned treatment.
8. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent form indicating voluntary consent to participate in the study prior to initiation of screening or study-related activities

General Exclusion Criteria:

1. History of major bleeding or clotting disorder
2. Females with a history of dysfunctional uterine bleeding
3. Smokers or use of tobacco and/or nicotine containing products within 3 months prior to dosing as determined by the subject's verbal history
4. Pregnant or breast-feeding
5. Males with a history of hormone therapy within 3 months prior to screening
6. Taking any type of chronic medication (including vitamin, nutritional and herbal supplements) for more than 14 consecutive days within the 4 weeks prior to study entry (use of hormonal contraceptives is acceptable)
7. Positive serologic test for human immunodeficiency virus (HIV), Hepatitis C virus antibody (HCV-Ab), or Hepatitis B surface antigen (HBsAg)
8. Donation of blood or blood products within 56 days prior to screening
9. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
10. Active drug or alcohol dependence within the prior 12 months or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services Inc., Secaucus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One study site in the US enrolled subjects between May 2017 and November 2019
Pre-assignment Details: 69 subjects enrolled; 64 subjects were randomized and 5 subjects were not randomized. Of the 5 subjects not randomized, 2 did not achieve a sufficient level of anticoagulation per protocol, 1 was withdrawn by Investigator decision (due to an asymptomatic low heart rate), 1 subject withdrew consent, and 1 had an AE during the rivaroxaban administration period causing discontinuation (T wave inversion observed on ECG).
Groups:
- Placebo: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of saline for injection (placebo) was administered.
- Ciraparantag 30mg: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of 30 mg ciraparantag was administered.
- Ciraparantag 60 mg: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of 60 mg ciraparantag was administered.
- Ciraparantag 120 mg: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of 120 mg ciraparantag was administered.
- Ciraparantag 180 mg: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of 180 mg ciraparantag was administered.
Period: Overall Study
Arm/Group | Placebo | Ciraparantag 30mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Ciraparantag 180 mg
Started | 16 | 12 | 12 | 12 | 12
Completed | 16 | 12 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 69 subjects were enrolled, and all of these subjects received at least 1 dose of rivaroxaban. Of these 69 subjects, 5 were not randomized, did not receive study drug (ciraparantag or placebo), and were discontinued from the study.
Groups:
- Ciraparantag 30 mg: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1-3. On Day 3, approximately 4 hours after last rivaroxaban dose, a single IV dose of 30 mg ciraparantag was administered.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Ciraparantag 180 mg | Total
Number analyzed (Participants) | 16 | 12 | 12 | 12 | 12 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (3.89) | 57.8 (5.67) | 56.1 (6.73) | 53.8 (3.10) | 55.9 (4.89) | 55.5 (5.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 0 | 3 | 9
  Male | 14 | 10 | 10 | 12 | 9 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 6 | 6 | 7 | 5 | 32
  Black or African American | 8 | 6 | 6 | 5 | 5 | 30
  Asian | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 12 | 12 | 12 | 12 | 64
Baseline Whole Blood Clotting Time (WBCT, manual method) [Mean (Standard Deviation); unit: minutes] | 7.8 (0.36) | 8.1 (0.42) | 7.8 (0.25) | 7.8 (0.33) | 7.9 (0.36) | 7.9 (.34)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Achieving Complete Reversal of Anticoagulation (WBCT is ≤ 110% of Baseline)
Description: Complete reversal is achieved if WBCT (manual method) is ≤ 110% of baseline at any post-baseline time point up to and including 1 hour following ciraparantag/placebo administration)
Time Frame: Within 1 Hour
Population: Pharmacodynamic population: all subjects who receive administration of study drug and provide at least one on-treatment whole blood clotting time measurement without protocol deviations with potential to affect these measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Ciraparantag 180 mg
Number analyzed (Participants) | 16 | 12 | 12 | 12 | 12
Participants | 3 | 7 | 11 | 11 | 12

2. Primary Outcome: Subjects Achieving Complete and Sustained Reversal of Anticoagulation (WBCT is ≤115%of Baseline)
Description: Complete and sustained reversal of anticoagulation is achieved for a subject if WBCT (manual method) is ≤ 115% of baseline at all time points between 1 and 8 hours (inclusive) following ciraparantag/placebo administration.
Time Frame: Between 1 and 8 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Ciraparantag 180 mg
Number analyzed (Participants) | 16 | 12 | 12 | 12 | 12
Participants | 3 | 8 | 11 | 11 | 12

ADVERSE EVENTS:
Time Frame: All AEs occurring after the subject signed the informed consent through the last study visit 7 to 10 days following ciraparantag/PBO administration). SAEs occurring up to 30 calendar days post treatment were collected.
Groups:
- Enrolled Not Randomized: Subjects received 20 mg rivaroxaban once daily in the morning on Days 1 up to Day 3. Subjects were not randomized and discontinued the study early (prior to treatment with ciraparantag) due to PI decision, subject withdraw, AE, or WBCT did not meet required threshold.
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Ciraparantag 180 mg | Enrolled Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12 | 0/12 | 0/12 | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12 | 0/12 | 0/12 | 1/12 | 0/5
Other Adverse Events (participants affected / at risk) | 3/16 | 0/12 | 2/12 | 8/12 | 10/12 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Ciraparantag 30 mg (N=12) | Ciraparantag 60 mg (N=12) | Ciraparantag 120 mg (N=12) | Ciraparantag 180 mg (N=12) | Enrolled Not Randomized (N=5)
Supraventricular Tachycardia (Cardiac disorders) | NA | NA | NA | NA | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Ciraparantag 30 mg (N=12) | Ciraparantag 60 mg (N=12) | Ciraparantag 120 mg (N=12) | Ciraparantag 180 mg (N=12) | Enrolled Not Randomized (N=5)
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 4 | 5 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 1 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03172910/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03172910/SAP_001.pdf